CLINICAL TRIAL: NCT03947099
Title: Ketamine Infusion Therapy for the Treatment of PTSD in Paramedics
Status: Completed | Type: Observational
Sponsor: Klarisana Physician Services PLLC (Industry)
Responsible Party: Sponsor
Other Study IDs: KRP002
Record Dates: First submitted 2019-05-08; First posted 2019-05-13 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Stress Disorders, Post-Traumatic; Anxiety Disorders
Keywords: ketamine; ptsd; depression; prehospital
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Depression | interventions — Ketamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Ketamine Hydrochloride — Participants are treated with six one-hour infusions of ketamine hydrochloride over a three week period in hopes of treating symptoms of PTSD.

SUMMARY:
This is an observational study to assess the change in several psychological screening tools before and after a series of six ketamine infusions in paramedics who suffer from post traumatic stress disorder as a result of working in emergency medical services.

DETAILED DESCRIPTION:
Working as a paramedic in a prehospital emergency medical services system (EMS) has been shown to lead to increased incidence of post traumatic stress disorder (PTSD) and increased risk of suicide in prehospital personnel. In recent years a growing body of literature has shown that ketamine hydrochloride can be an effective treatment for PTSD. This study seeks to look specifically at paramedic level emergency medical technicians ("paramedics") with PTSD related to their prehospital work and assess whether ketamine infusion therapy can be an effective treatment for them. This is an observational study where the results of psychological screening tools that are administered before and after a six-infusion series are reported. Additionally the same assessment tools will be administered again 30 days after the final treatment to measure the durability of any changes. The participants will receive the Periodic Health Questionnaire-9 (PHQ-9), the PTSD Checklist for Diagnostic and Statistical Manual, DSM-5 (PCL-5), the Alcohol Use Disorders Identification Test (AUDIT), and the Beck Anxiety Inventory (BAI) before the infusions, after the series of six, and thirty days later. Additionally, after the series of six infusions, participants will receive the Revised Mystical Experience Questionnaire-30 (RMEQ-30) and a one question survey to assess the impact of the experiential aspect of ketamine.

ELIGIBILITY:
Inclusion Criteria:

* Must have worked as a paramedic (EMT-P) on a 911 prehospital service for at least five years.
* Must be diagnosed with post traumatic stress disorder that happened as a result of working as a paramedic
* Diagnosis must have been made by a mental health professional
* The symptoms of PTSD must be having a significant adverse effect on the subject's life
* Subjects must be able to speak and read English

Exclusion Criteria:

* Currently participating in another PTSD treatment program and/or research study
* Diagnosis of psychosis
* Uncontrolled hypertension or a history of heart failure

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Men and women who are trained as paramedics (EMT-P) and have worked in 911 emergency medical service systems for at least five years.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-02-22 (Actual)

PRIMARY OUTCOMES:
PHQ-9 Score to assess for symptoms of depression | three weeks
  Assess for an improvement in the Periodic Health Questionnaire nine (PHQ-9) score after a series of six ketamine infusions. The PHQ-9 is a nine question scale followed by a single question that assesses functional impairment. Each of the nine questions are scored on a basis of zero to four. The higher the score the more severe the symptoms of depression are. The highest score is 27 and the lowest is zero.
PCL-5 Score to assess for symptoms of PTSD | three weeks
  Assess for an improvement in the PTSD Checklist for Diagnostic and Statistical Manual version five (PCL-5) score after a series of six ketamine infusions. The PCL-5 is a 20 question scale and each question is scored on a zero to four scale. A higher score indicates more severe symptoms of PTSD. The highest score possible is 80 and the lowest is zero.

SECONDARY OUTCOMES:
Assessment of the experiential impact of ketamine therapy | three weeks
  The investigators seek to determine the role that the experiential (psychedelic) aspect of ketamine plays in the treatment of PTSD. This will utilize the Mystical Experience Questionnaire 30. This is a 30 question screening instrument where each question is scored on a scale of one to five. The maximum score is 150. A higher score indicates that the participant reports a more powerful mystical experience. There is also a single question that asks the participants to rate on a scale of one to five how important they feel the experiential (or psychedelic) aspect of the therapy was to their treatment. Five would indicate that they felt it was an important part of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Carl J Bonnett, MD, Principal Investigator — Klarisana Physician Services PLLC
Locations (1):
- Klarisana, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Luftman K, Aydelotte J, Rix K, Ali S, Houck K, Coopwood TB, Teixeira P, Eastman A, Eastridge B, Brown CV, Davis M. PTSD in those who care for the injured. Injury. 2017 Feb;48(2):293-296. doi: 10.1016/j.injury.2016.11.001. Epub 2016 Nov 10. PMID 27871770
- [Result] Jacobowitz W. PTSD in psychiatric nurses and other mental health providers: a review of the literature. Issues Ment Health Nurs. 2013 Nov;34(11):787-95. doi: 10.3109/01612840.2013.824053. PMID 24131410
- [Result] Stanley IH, Hom MA, Joiner TE. Suicide mortality among firefighters: Results from a large, urban fire department. Am J Ind Med. 2016 Nov;59(11):942-947. doi: 10.1002/ajim.22587. Epub 2016 May 24. PMID 27219513
- [Result] Bing-Canar H, Ranney RM, McNett S, Tran JK, Berenz EC, Vujanovic AA. Alcohol Use Problems, Posttraumatic Stress Disorder, and Suicide Risk Among Trauma-Exposed Firefighters. J Nerv Ment Dis. 2019 Mar;207(3):192-198. doi: 10.1097/NMD.0000000000000947. PMID 30724832
- [Result] Abdallah CG, Roache JD, Averill LA, Young-McCaughan S, Martini B, Gueorguieva R, Amoroso T, Southwick SM, Guthmiller K, Lopez-Roca AL, Lautenschlager K, Mintz J, Litz BT, Williamson DE, Keane TM, Peterson AL, Krystal JH; Consortium to Alleviate PTSD. Repeated ketamine infusions for antidepressant-resistant PTSD: Methods of a multicenter, randomized, placebo-controlled clinical trial. Contemp Clin Trials. 2019 Jun;81:11-18. doi: 10.1016/j.cct.2019.04.009. Epub 2019 Apr 15. PMID 30999057
- See also: The sponsoring treatment facility for this study — http://www.klarisana.com